CLINICAL TRIAL: NCT02424799
Title: A Randomised Double Blind (Sponsor Unblinded), Single and Repeat Ascending Dose First Time in Human Study in Healthy Subjects, Cold Urticaria and Chronic Spontaneous Urticaria Subjects to Investigate Safety, Tolerability, Pharmacodynamics and Pharmacokinetics of GSK2646264
Brief Title: Study to Investigate Safety, Tolerability, Pharmacodynamics and Pharmacokinetics of GSK2646264
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 200196; 2014-001015-39 (EudraCT Number)
Record Dates: First submitted 2014-11-13; First posted 2015-04-23 (Estimated); Results first posted 2019-06-21 (Actual); Last update posted 2019-06-21 (Actual); Status verified 2019-03

CONDITIONS: Urticaria
Keywords: Urticaria; SYK Inhibitor
MeSH Terms: conditions — Urticaria | interventions — GSK2646264

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- Part A: Dose group 1 (Experimental): Subjects will be treated topically with 0.5 % GSK2646264 cream and placebo cream on an area of approximately 12 x 3 centimetre (cm) on the volar aspect of the arm which approximates to 0.2% total body surface area (BSA), on each arm. On Day 2 and Day 3 subjects will receive active treatment and placebo on the same arms as on Day 1, with the percentage BSA being 1% on Day 2 and 5% on Day 3.
  Interventions: Drug: GSK2646264 0.5% topical cream; Drug: Placebo
- Part A: Dose group 2 (Experimental): Subjects will be treated topically with 1 % GSK2646264 cream and placebo cream on the morning and evening of Day 1 starting at the final % BSA dosed at Day 3 in group 1 which is anticipated to be 5%. In dose group 2, the starting BSA will increase to 10% at Day 3 and then 20% by Day 5. Administration of the evening (PM) dose will be dependent on the data from Part A Dose group 1.
  Interventions: Drug: GSK2646264 0.5% topical cream; Drug: GSK2646264 1% topical cream; Drug: Placebo
- Part B (Experimental): Cold urticaria subjects will receive treatment to 4 defined areas (right and left arms and legs). Subjects will be treated with maximum tolerated strength of GSK2646264 cream (0.5% or 1%) and placebo cream in morning or in morning and evening to 2 specified areas of ~5% BSA on the subject's legs for the CU assessment and to 2 specified areas of 0.2% BSA on the volar aspect of the arm. The maximum tolerated strength and evening dosing will be dependent on the data from the Part A
  Interventions: Drug: GSK2646264 0.5% topical cream; Drug: GSK2646264 1% topical cream; Drug: Placebo
- Part C (Experimental): Chronic spontaneous urticaria subjects will be treated with the maximum tolerated strength of GSK2646264 cream from Part A (0.5% or 1%) and placebo cream onto defined areas (right and left arms and, legs and front torso) from Days 1 to 7. The total % BSA for an individual subject will be decided by the investigator prior to randomization. The maximum % BSA and the frequency of dosing will be decided after part A of the study.
  Interventions: Drug: GSK2646264 0.5% topical cream; Drug: GSK2646264 1% topical cream; Drug: Placebo

INTERVENTIONS:
Drug: GSK2646264 0.5% topical cream — GSK2646264 0.5% topical cream is supplied as white-to-off-white aqueous cream stored in amber glass jars
Drug: GSK2646264 1% topical cream — GSK2646264 1% topical cream is supplied as white-to-off-white aqueous cream stored in amber glass jars
  Arms: Part A: Dose group 2; Part B; Part C
Drug: Placebo — Placebo topical cream is supplied as white-to-off-white aqueous cream stored in amber glass jars

SUMMARY:
This First Time in Human (FTIH) study, which will be performed in three parts, is designed to investigate the safety, local tolerability, pharmacokinetics and pharmacodynamics after single and repeat topical applications of up to 2 strengths of GSK2646264 and corresponding placebo within the same subject, in healthy adult subjects (Part A), subjects with cold urticaria (CU, Part B) and subjects with chronic spontaneous urticaria (CsU, Part C). The study will also measure short term effects of GSK2646264 on the number and size of weals in subjects with CsU, and in healthy subjects and subjects with CU following provocation tests.

ELIGIBILITY:
Inclusion criteria for all subjects in Parts A, B and C

* Male or female subject aged at least 18 years (Yrs) at the time of signing the informed consent. The upper age limit of subjects is defined in the specific inclusion criteria for each cohort.
* All subjects must be free from scarring or skin markings (e.g. tattoos or piercings) and open wounds (e.g. scarring or skin markings) on the defined areas of the body that cream will be applied onto, unless in the opinion of the investigator it will not compromise the subjects safety and quality of data.
* Able to refrain from exposure to extended and direct sunlight during the study period, from screening (SCR) until follow up, especially the area that is under treatment during the study.
* Able to refrain from shaving and waxing the areas on which the study cream will be applied during the duration of the study from SCR to follow up.
* Male subjects with female partners of child-bearing potential must agree to use one of the contraception methods listed in protocol. This criterion must be followed from the time of the first dose of study medication until the follow up visit or a time period that is 5 terminal half-live post-last dose which will be determined following Part A of the study.
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form. Willing, committed and able to return for all clinic visits and complete all study-related procedures. Able to read, understand and complete study- related questionnaires.

Inclusion criteria specific for healthy subjects (Part A)

* The subject is aged between 18 and 55 yrs of age inclusive, at the time of signing the informed consent.
* Body weight >=50 kilogram (kg) and body mass index (BMI) within the range 19 to 30 kg per square meter (m^2 )(inclusive).
* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring. A subject with a clinical abnormality or laboratory parameter(s) which is/are not specifically listed in the inclusion or exclusion criteria, outside the reference range for the population being studied may be included only if the Investigator, in consultation with the GSK Medical Monitor (MM) if required, agrees and documents that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Demonstration of a positive weal and flare reaction (>=3 millimeter (mm) in diameter relative to negative control) to at least one allergen from a battery of allergens (mixed grass pollen, Dermatophagoides pteronyssinus, birch pollen and cat dander) on skin prick testing at SCR.
* Subjects must be free from any past or present benign or malignant skin conditions and disease, unless in the opinion of the investigator it will not compromise the subject's safety and quality of data.
* Non-smokers or if the subject is a tobacco smoke: smokes less than 5 cigarettes per day and commits to not smoke tobacco for the duration of the in-house stay, and commits to stable and moderate use (as determined by the Investigator) of tobacco or nicotine-containing products, including nicotine patches/gum, during the course of the study, as long as the patches do not interfere with the study procedures.
* A female subject is eligible to participate if she is of: Non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy for this definition, "documented" refers to the outcome of the investigator's/designee's review of the subject's medical history for study eligibility, as obtained via a verbal interview with the subject or from the subject's medical records; or postmenopausal defined as 12 months of spontaneous amenorrhea in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) >40 milli international unit [MlU]/milliliter [mL] and estradiol <40 picogram (pg)/mL (<147 picomoles/litre) is confirmatory. Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the contraception methods described if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrolment. For most forms of HRT, at least 2-4 weeks will elapse between the cessation of therapy and the blood draw; this interval depends on the type and dosage of HRT. Following confirmation of their post-menopausal status, they can resume use of HRT during the study without use of a contraceptive method.

Additional Inclusion criteria specific for subjects with CU (Part B)

* Diagnosed with CU for more than six weeks as confirmed by medical history and with a positive cold stimulation test assessed by TEMPTest 4.0 prior to first dose.
* The subject is aged between 18 and 70 yrs of age inclusive, at the time of signing the informed consent.
* Body weight >=50 kg and BMI within the range 19 to 35 kg/m^2 (inclusive).
* Other than a diagnosis of CU, the subject should have no other co-morbidities which would introduce additional risk factors and will not interfere with the study procedures, as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring.
* A subject with a clinical abnormality or laboratory parameter(s) which is/are not specifically listed in the inclusion or exclusion criteria, outside the reference range for the population being studied may be included only if the Investigator, in consultation with the GSK MM if required, agrees and documents that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedure.
* In addition, the following criterion will apply to a minimum of 4 patients in Part B: Demonstration of a positive weal and flare reaction (>=3 mm relative to negative control) to at least one allergen from a battery of allergens (mixed grass pollen, Dermatophagoides pteronyssinus, birch pollen and cat dander) on skin prick testing at SCR,
* Subjects must be free from any past or present benign or malignant skin conditions and disease, other than the specified condition required for eligibility of subjects as defined in the specific inclusion criteria for CU cohort unless in the opinion of the investigator it will not compromise the subjects safety and quality of data.
* Non-smokers or if the subject is a tobacco smoker: smokes less than 5 cigarettes per day and commits to not smoke tobacco for the duration of the in-house stay, and commits to stable and moderate use (as determined by the Investigator) of tobacco or nicotine-containing products, including nicotine patches/gum, during the course of the study, as long as the patches do not interfere with the study procedures.
* Female subjects must agree to use one of the contraception methods listed in protocol, 28 days before their SCR visit and until the followup visit or a time period that is 5 terminal half-live post-last dose which will be determined following Part A of the study.

Additional Inclusion criteria specific for subjects with CsU (Part C)

* The subject is aged between 18 and 70 yrs of age inclusive, at the time of signing the informed consent.
* Body weight >=50 kg and BMI within the range 19 to 35 kg/m2 (inclusive)
* Subjects who have a score of >14 on the UAS7 questionnaire with between 4-10 weals observed in a defined area of the body will be included in this study. This area must include either both arms, or both legs or both sides of their torso for 7 consecutive days during the SCR period, prior to the Day 1 visit. If a subject has not completed 7 consecutive days of UAS questionnaire prior to dosing on Day 1 due to exceptional circumstances, the SCR period may be extended until the subject has completed 7 consecutive days of UAS questionnaire. This will only be at the discretion of the Investigator.
* No other aetiology identified for chronic urticaria such as drug-related or inducible urticaria as determined by history, physical examination and laboratory studies.
* Subjects must be free from any past or present benign or malignant skin conditions and disease, other than the specified condition required for eligibility of subjects as defined in the specific inclusion criteria for CsU cohort unless in the opinion of the investigator it will not compromise the subjects safety and quality of data.
* Other than a diagnosis of CsU the subject should have no other co-morbidities which would introduce additional risk factors and will not interfere with the study procedures, as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring.
* A subject with a clinical abnormality or laboratory parameter(s) which is/are not specifically listed in the inclusion or exclusion criteria, outside the reference range for the population being studied may be included only if the Investigator, in consultation with the GSK MM if required, agrees and documents that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Female subjects must agree to use one of the contraception methods 28 days before their SCR visit listed in protocol and until the follow-up visit or a time period that is 5 terminal half-live post-last dose which will be determined following Part A of the study.

All Cohorts Exclusion Criteria

* Thyroid stimulating hormone levels outside normal range.
* Subjects with a history of Graves disease.
* Subjects with a history of any thyroid cancer.
* Unable or unwilling to avoid use of topical creams/lotions at sites where medication will be applied. Washing with soap and water will be permitted.
* Based on averaged corrected QT interval for heart rate (Fridericia's) [QTcF] values of triplicate ECGs obtained over a brief recording period: QTcF > 450 msec; or QTcF >480 milliseconds (msec) in subjects with Bundle Branch Block.
* Alanine aminotransferase, alkaline phosphatase and bilirubin ≥ 1.5x upper limit of normal (ULN) (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones) or previous history of uncomplicated cholecystectomy.
* History of regular alcohol consumption within 6 months of the study defined as: An average weekly intake of >21 units for males or >14 units for females. One unit is equivalent to 8 g of alcohol: a half-pint (~240 mL) of beer, 1 glass (125 mL) of wine or 1 (25 mL) measure of spirits.
* History of sensitivity to any of the study medications, or components thereof, history of anaphylaxis or a history of drug or other allergy that, in the opinion of the investigator or GSK MM, contraindicates their participation.
* Unable to refrain from vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half lives (whichever is longer) prior to the SCR visit until the completion of the follow-up assessments, unless in the opinion of the Investigator, in consultation with the GSK MM if required, the medication will not interfere with the study procedures or compromise subject safety.
* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of SCR.
* A positive test for HIV antibody.
* Lactating females.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day
* Use of topical steroids or calcinurin inhibitors are prohibited during the study from SCR to follow up.
* Exclusion related to prior drug treatments: Intake of oral corticosteroids within 7 days >10 milligram (mg) per day prior to first SCR visit; Use of depot corticosteroids within 7 days prior to first SCR visit; Subjects who are taking anticoagulants (e.g. warfarin) must not be on warfarin within 21 days prior to SCR. Subjects who are having psoralen combined with ultraviolet A (PUVA) treatment must not be using PUVA treatment within 21 days prior to SCR.
* Subjects who work for the Sponsor, CRO, or one of the study centres. Country Specific Exclusion criteria for Germany that applies to Part A, Part B and Part C.
* Subjects who live in detention on court order or on regulatory action, see §40 subsection 1 sentence 3 no. 4 AMG. (Arzneimittelgesetz).

Additional Exclusion for Part A - Healthy Subjects

* Use of H1 antihistamines within 3 days prior to first SCR visit Additional Exclusion for Part B - CU Subjects
* Exclusion related to prior drug treatments: Use of Zaditen (Ketotifen) within 14 days prior to first SCR visit; Use of Doxepin AZU and other tricyclic antidepressants with antihistaminergic properties within 14 days prior to first SCR visit; Use of H2 antihistamines within 7 days prior to first SCR visit; Use of H1 antihistamines within 7 days prior to first SCR visit; Use of monteleukast or any other leukotriene antagonist within 7 days prior to first SCR visit; Use of biologicals including omalizumab within 5 months prior to first SCR visit.

Additional Exclusion for Part C- CsUpatients

* Exclusion related to prior drug treatments: Intake of cyclosporin within 10 days prior to first SCR visit; Intake of other immunosuppressant drugs within 28 days of first SCR visit; Use of monteleukast or any other leukotriene antagonist within 7 days prior to first SCR visit; Use of Dapsone within 7 days prior to first SCR visit; Use of Zaditen (Ketotifen) within 14 days prior to first SCR visit; Use of Doxepin AZU and other tricyclic antidepressants with antihistaminergic properties within 14 days prior to first SCR visit; Use of H2 antihistamines within 7 days prior first SCR visit; Use of biologicals including omalizumab within 5 months prior to first SCR visit; Use of H1 antihistamines above the licensed dose within 3 days prior to first SCR visit.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2014-11-17 (Actual); Primary Completion 2017-11-10 (Actual); Study Completion 2017-11-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline; GSK Clinical Trials, Study Director — GlaxoSmithKline (for GlaxoSmithKline; Human Genome Sciences Inc., a GSK Company; Sirtris, a GSK Company; Stiefel, a GSK Company; ViiV Healthcare)
Locations (3):
- GSK Investigational Site, Berlin, Germany
- United Kingdom (2):
  - GSK Investigational Site, Norwich, Norfolk
  - GSK Investigational Site, London

REFERENCES:
- [Derived] Dickson MC, Walker A, Grattan C, Perry H, Williams N, Ratia N, Dewit O, Gisbert S, Metz M, Maurer M. Effects of a topical treatment with spleen tyrosine kinase inhibitor in healthy subjects and patients with cold urticaria or chronic spontaneous urticaria: Results of a phase 1a/b randomised double-blind placebo-controlled study. Br J Clin Pharmacol. 2021 Dec;87(12):4797-4808. doi: 10.1111/bcp.14923. Epub 2021 Jun 18. PMID 34020509

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted from 17-November-2014 to 10-November-2017 at centers two centers in the United Kingdom and two centers in Germany.
Pre-assignment Details: 92 participants were screened (3 re-screened) of which 58 were screen failures. Hence 34 participants, 17 healthy participants (Part A), 12 participants with cold urticaria (CU, Part B) and 5 participants with chronic spontaneous urticaria (CsU, Part C) were randomized.
Groups:
- Part A-GSK2646264 0.5% and Placebo: Participants were treated topically with 0.5 % GSK2646264 cream and placebo cream on an area of approximately 12 x 3 centimeter (cm) on the volar aspect of the arm which approximated to 0.2% total body surface area (BSA), on each arm. On Day 2 and Day 3 participants received active treatment and placebo on the same arms as on Day 1, with the percentage BSA being 1% on Day 2 and 5% on Day 3.
- Part A-GSK2646264 1% and Placebo: Participants received active treatment (1% cream strength) and placebo on Days 1, 2, 3 and 4. On Day 1 and Day 2, participants received treatment to 0.2% BSA; active treatment on one arm and placebo on the other arm. In addition, participants received treatment to another 5% BSA; active to one side of the torso and placebo to the other. On Days 3 and 4, the same treatment to the arms was applied as on Days 1 and 2, but the %BSA of the torso to which treatment was applied to was increased to 10%.
- Part B-Placebo: CU participants received matching placebo treatment to an area of 10% BSA (5% BSA on each arm, n=1) or 3.5% BSA (spread over the 2 arms, n=2) on Days 1, 2 and 3
- Part B GSK2646264 1%: CU participants received 1% strength GSK2646264 to an area of 10% BSA (5% BSA on each arm, n=3) or 3% BSA (spread over the 2 arms, n=6) on Days 1, 2 and 3
- Part C-Placebo: CSU participants received matching placebo treatment to 10% BSA (arms, legs or torso) on Days 1, 4 and 7.
- Part C GSK2646264 1%: CSU participants received 1% strength GSK2646264 to 10% BSA (arms, legs or torso) on Days 1, 4 and 7.
Period: Part A (Up to Day 11)
Arm/Group | Part A-GSK2646264 0.5% and Placebo | Part A-GSK2646264 1% and Placebo | Part B-Placebo | Part B GSK2646264 1% | Part C-Placebo | Part C GSK2646264 1%
Started | 9 | 8 | 0 | 0 | 0 | 0
Completed | 9 | 8 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Part B (Up to Day 19)
Arm/Group | Part A-GSK2646264 0.5% and Placebo | Part A-GSK2646264 1% and Placebo | Part B-Placebo | Part B GSK2646264 1% | Part C-Placebo | Part C GSK2646264 1%
Started | 0 | 0 | 3 | 9 | 0 | 0
Completed | 0 | 0 | 3 | 9 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Part C (Up to Day 23)
Arm/Group | Part A-GSK2646264 0.5% and Placebo | Part A-GSK2646264 1% and Placebo | Part B-Placebo | Part B GSK2646264 1% | Part C-Placebo | Part C GSK2646264 1%
Started | 0 | 0 | 0 | 0 | 1 | 4
Completed | 0 | 0 | 0 | 0 | 1 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Part A-GSK2646264 0.5% and Placebo: Participants were treated topically with 0.5 % GSK2646264 cream and placebo cream on an area of approximately 12 x 3 cm on the volar aspect of the arm which approximated to 0.2% total BSA, on each arm. On Day 2 and Day 3 participants received active treatment and placebo on the same arms as on Day 1, with the percentage BSA being 1% on Day 2 and 5% on Day 3.
- Total: Total of all reporting groups
Arm/Group | Part A-GSK2646264 0.5% and Placebo | Part A-GSK2646264 1% and Placebo | Part B-Placebo | Part B GSK2646264 1% | Part C-Placebo | Part C GSK2646264 1% | Total
Number analyzed (Participants) | 9 | 8 | 3 | 9 | 1 | 4 | 34
Age, Continuous [Mean (Standard Deviation); unit: Years] | 38.0 (10.74) | 38.9 (11.54) | 41.3 (10.07) | 50.7 (11.70) | 24.0 (NA) — Standard deviation could not be calculated as a single participant was analyzed. | 50.8 (12.58) | 42.9 (12.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 2 | 7 | 1 | 4 | 17
  Male | 7 | 7 | 1 | 2 | 0 | 0 | 17
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White/Caucasian/European Heritage | 9 | 8 | 3 | 8 | 0 | 4 | 32
  White-Arabic/North African Heritage | 0 | 0 | 0 | 1 | 1 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs) and Serious AEs (SAEs) Part A
Description: AE is any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An SAE is any untoward medical occurrence that, at any dose results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, or is a congenital anomaly/birth defect or is medically significant. Safety population comprised of all participants who took at least one dose of study treatment.
Time Frame: Up to Day 7
Population: Safety Population
Measure: Count of Participants; unit: Participants
Groups:
- Part A-GSK2646264 0.5%: Participants were treated topically with 0.5 % GSK2646264 cream and placebo cream on an area of approximately 12 x 3 cm on the volar aspect of the arm which approximated to 0.2% total BSA, on each arm. On Day 2 and Day 3 participants received active treatment and placebo on the same arms as on Day 1, with the percentage BSA being 1% on Day 2 and 5% on Day 3.
Arm/Group | Part A-GSK2646264 0.5%
Number analyzed (Participants) | 9
Participants
  AEs | 4
  SAEs | 0

2. Primary Outcome: Number of Participants With AEs and SAEs Part A
Description: AE is any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An SAE is any untoward medical occurrence that, at any dose results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, or is a congenital anomaly/birth defect or is medically significant.
Time Frame: Up to Day 11
Population: Safety Population
Measure: Count of Participants; unit: Participants
Groups:
- Part A-GSK2646264 1%: Participants received active treatment (1% cream strength) on Days 1, 2, 3 and 4. On Day 1 and Day 2, participants received treatment to 0.2% BSA; active treatment on one arm. In addition, participants received treatment to another 5% BSA; active to one side of the torso. On Days 3 and 4, the same treatment to the arms was applied as on Days 1 and 2, but the %BSA of the torso to which treatment was applied to was increased to 10%.
Arm/Group | Part A-GSK2646264 1%
Number analyzed (Participants) | 8
Participants
  AEs | 4
  SAEs | 0

3. Primary Outcome: Number of Participants With AEs and SAEs Part B
Description: AE is any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An SAE is any untoward medical occurrence that, at any dose results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, or is a congenital anomaly/birth defect or is medically significant. Data is presented according to the percentage BSA as it impacted safety
Time Frame: Up to Day 19
Population: Safety Population
Measure: Count of Participants; unit: Participants
Groups:
- Part B (10% BSA)-Placebo: CU participants received matching placebo treatment to an area of 10% BSA (5% BSA each arm) on Days 1, 2 and 3.
- Part B (10% BSA) GSK2646264 1%: CU participants received 1% strength GSK2646264 treatment to an area of 10% BSA (5% BSA on each arm) on Days 1, 2 and 3.
- Part B (3.5% BSA)-Placebo: CU participants received matching placebo treatment to an area of 3.5% BSA (spread over the 2 arms) on Days 1, 2 and 3.
- Part B (3.5% BSA) GSK2646264 1%: CU participants received 1% strength GSK2646264 treatment to an area of 3.5% BSA (spread over the 2 arms) on Days 1, 2 and 3.
Arm/Group | Part B (10% BSA)-Placebo | Part B (10% BSA) GSK2646264 1% | Part B (3.5% BSA)-Placebo | Part B (3.5% BSA) GSK2646264 1%
Number analyzed (Participants) | 1 | 3 | 2 | 6
Participants
  AEs | 1 | 3 | 0 | 3
  SAEs | 0 | 0 | 0 | 0

4. Primary Outcome: Number of Participants With AEs and SAEs Part C
Description: as for outcome 2
Time Frame: Up to Day 23
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part C-Placebo | Part C GSK2646264 1%
Number analyzed (Participants) | 1 | 4
Participants
  AEs | 1 | 1
  SAEs | 0 | 0

5. Primary Outcome: Number of Participants With AEs and SAEs Defined by Severity Part A
Description: AE is any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An SAE is any untoward medical occurrence that, at any dose results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, or is a congenital anomaly/birth defect or is medically significant. AE and SAE were categorized as mild=an event that was easily tolerated by the participant, causing minimal discomfort and not interfering with everyday activities, moderate=an event that was sufficiently discomforting to interfere with normal everyday activities and severe=an event that prevented normal everyday activities.
Time Frame: Up to Day 7
Population: Safety Population
Measure: Count of Participants; unit: Participants
Groups:
- Part A-GSK2646264 0.5%: Participants were treated topically with GSK2646264 0.5% cream on an area of approximately 12 x 3 cm on the volar aspect of the arm which approximated to 0.2% total BSA, on each arm. On Day 2 and Day 3 participants received active treatment and placebo on the same arms as on Day 1, with the percentage BSA being 1% on Day 2 and 5% on Day 3.
Arm/Group | Part A-GSK2646264 0.5%
Number analyzed (Participants) | 9
Participants
  Mild | 3
  Moderate | 1
  Severe | 0

6. Primary Outcome: Number of Participants With AEs and SAEs Defined by Severity Part A
Description: as for outcome 5
Time Frame: Up to Day 11
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part A-GSK2646264 1%
Number analyzed (Participants) | 8
Participants
  Mild | 3
  Moderate | 1
  Severe | 0

7. Primary Outcome: Number of Participants With AEs and SAEs Defined by Severity Part B
Description: AE is any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An SAE is any untoward medical occurrence that, at any dose results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, or is a congenital anomaly/birth defect or is medically significant. AE and SAE were categorized as mild=an event that was easily tolerated by the participant, causing minimal discomfort and not interfering with everyday activities, moderate=an event that was sufficiently discomforting to interfere with normal everyday activities and severe=an event that prevented normal everyday activities. Data is presented according to the percentage BSA as it impacted safety
Time Frame: Up to 19 days
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part B (10% BSA)-Placebo | Part B (10% BSA) GSK2646264 1% | Part B (3.5% BSA)-Placebo | Part B (3.5% BSA) GSK2646264 1%
Number analyzed (Participants) | 1 | 3 | 2 | 6
Participants
  Mild | 1 | 2 | 0 | 2
  Moderate | 0 | 1 | 0 | 1
  Severe | 0 | 0 | 0 | 0

8. Primary Outcome: Number of Participants With AEs and SAEs Defined by Severity Part C
Description: as for outcome 5
Time Frame: Up to 23 days
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part C-Placebo | Part C GSK2646264 1%
Number analyzed (Participants) | 1 | 4
Participants
  Mild | 1 | 1
  Moderate | 0 | 0
  Severe | 0 | 0

9. Primary Outcome: Change From Baseline in Vital Sign Parameter Heart Rate for Part A
Description: Vital sign heart rate was measured in the semi-supine position after 10 minutes of rest. Assessments were performed at Day 2, Day 3, Day 4 and follow-up. Baseline was defined as assessments performed at Day 1(pre-dose). Change from Baseline was calculated as the post-dose visit value minus the Baseline value.
Time Frame: Baseline (Day 1 pre-dose) and Day 2 (pre-dose), Day 3 (pre-dose), Day 4 and follow-up (Day 5 to Day 7)
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Beats/minute
Arm/Group | Part A-GSK2646264 0.5%
Number analyzed (Participants) | 9
Beats/minute
  Day 2 - Pre-dose | 0.2 (5.43)
  Day 3 - Pre-dose | 0.9 (6.01)
  Day 4 | 3.0 (7.12)
  Follow-up | 10.4 (9.32)

10. Primary Outcome: Change From Baseline in Vital Sign Parameter Heart Rate for Part A
Description: Vital sign heart rate was measured in the semi-supine position after 10 minutes of rest. Assessments were performed at Day 2 (pre-dose), Day 3 (pre-dose), Day 4 (pre-dose), Day 5, Day 6, Day 7, Day 8 and follow-up. Baseline was defined as assessments performed at Day 1(pre-dose). Change from Baseline was calculated as the post-dose visit value minus the Baseline value.
Time Frame: Baseline (Day 1 pre-dose) and Day 2 (pre-dose), Day 3 (pre-dose), Day 4 (pre-dose), Day 5, Day 6, Day 7, Day 8 and follow-up (Day 9 to Day 11)
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Beats/minute
Arm/Group | Part A-GSK2646264 1%
Number analyzed (Participants) | 8
Beats/minute
  Day 2 - Pre-dose | -2.1 (5.99)
  Day 3 - Pre-dose | 1.0 (5.53)
  Day 4 - Pre-dose | -0.8 (5.50)
  Day 5 | -1.9 (3.91)
  Day 6 | 1.0 (2.51)
  Day 7 | 2.0 (4.07)
  Day 8 | 3.9 (4.61)
  Follow-up | 8.0 (8.73)

11. Primary Outcome: Change From Baseline in Vital Sign Parameter Heart Rate for Part B
Description: Vital sign heart rate was measured in the semi-supine position after 10 minutes of rest. Assessments were performed at Day 2 (pre-dose), Day 3 (pre-dose), Day 6, Day 9, Day 12, Day 15 and follow-up. Baseline was defined as assessments performed at Day 1(pre-dose). Change from Baseline was calculated as the post-dose visit value minus the Baseline value.
Time Frame: Baseline (Day 1 pre-dose) and Day 2 (pre-dose), Day 3 (pre-dose), Day 6, Day 9, Day 12, Day 15 and follow-up (Day 17 to Day 19)
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Beats/minute
Arm/Group | Part B-Placebo | Part B GSK2646264 1%
Number analyzed (Participants) | 3 | 9
Beats/minute
  Day 2 - Pre-dose | 8.0 (6.93) | -1.1 (8.07)
  Day 3 - Pre-dose | 10.0 (5.29) | -0.9 (10.73)
  Day 6 | 4.0 (4.0) | 2.9 (16.10)
  Day 9 | 14.0 (3.46) | 2.6 (13.39)
  Day 12 | 16.0 (10.58) | 8.0 (14.70)
  Day 15 | 19.3 (11.02) | 4.9 (17.41)
  Follow-up | 12.0 (13.86) | 2.0 (18.44)

12. Primary Outcome: Change From Baseline in Vital Sign Parameter Heart Rate for Part C
Description: Vital sign heart rate was measured in the semi-supine position after 10 minutes of rest. Assessments were performed at Day 4 (pre-dose), Day 7 (pre-dose), Day 10, Day 15 and follow-up. Baseline was defined as assessments performed at Day 1(pre-dose). Change from Baseline was calculated as the post-dose visit value minus the Baseline value. NA indicates standard deviation could not be calculated as a single participant was analyzed.
Time Frame: Baseline and (Day 1 pre-dose), Day 4 (pre-dose), Day 7 (pre-dose), Day 10, Day 15, follow-up (Day 23)
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Beats/minute
Arm/Group | Part C-Placebo | Part C GSK2646264 1%
Number analyzed (Participants) | 1 | 4
Beats/minute
  Day 4 - Pre-dose | 16.0 (NA) — NA indicates standard deviation could not be calculated as a single participant was analyzed. | 4.8 (3.95)
  Day 7 - Pre-dose | 4.0 (NA) — NA indicates standard deviation could not be calculated as a single participant was analyzed. | 2.3 (5.56)
  Day 10 | 20.0 (NA) — NA indicates standard deviation could not be calculated as a single participant was analyzed. | 8.5 (7.72)
  Day 15 | 20.0 (NA) — NA indicates standard deviation could not be calculated as a single participant was analyzed. | 14.3 (5.06)
  Follow-up | 8.0 (NA) — NA indicates standard deviation could not be calculated as a single participant was analyzed. | 6.0 (6.73)

13. Primary Outcome: Change From Baseline in Vital Sign Parameters Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP) for Part A
Description: Vital signs SBP and DBP were measured in the semi-supine position after 10 minutes of rest. Assessments were performed at Day 2, Day 3, Day 4 and follow-up. Baseline was defined as assessments performed at Day 1 (pre-dose). Change from Baseline was calculated as the post-dose visit value minus the Baseline value.
Time Frame: Baseline (Day 1 pre-dose) and Day 2 (pre-dose), Day 3 (pre-dose), Day 4 and follow-up (Day 5 to Day 7)
Measure: Mean (Standard Deviation); unit: millimeters of mercury
Arm/Group | Part A-GSK2646264 0.5%
Number analyzed (Participants) | 9
millimeters of mercury
  SBP, Day 2 - Pre-dose | -0.1 (11.21)
  SBP, Day 3 - Pre-dose | -0.9 (7.27)
  SBP, Day 4 | -1.1 (9.31)
  SBP, Follow-up | 4.1 (11.38)
  DBP, Day 2 - Pre-dose | -0.3 (4.50)
  DBP, Day 3 - Pre-dose | 0.6 (6.52)
  DBP, Day 4 | 2.2 (4.29)
  DBP, Follow-up | 4.2 (6.85)

14. Primary Outcome: Change From Baseline in Vital Sign Parameters SBP and DBP for Part A
Description: Vital signs SBP and DBP were measured in the semi-supine position after 10 minutes of rest. Assessments were performed at Day 2 (pre-dose), Day 3 (pre-dose), Day 4 (pre-dose), Day 5, Day 6, Day 7, Day 8 and follow-up. Baseline was defined as assessments performed at Day 1 (pre-dose). Change from Baseline was calculated as the post-dose visit value minus the Baseline value.
Time Frame: as for outcome 10
Population: Safety Population
Measure: Mean (Standard Deviation); unit: millimeters of mercury
Arm/Group | Part A-GSK2646264 1%
Number analyzed (Participants) | 8
millimeters of mercury
  SBP, Day 2 - Pre-dose | 1.0 (12.41)
  SBP, Day 3 - Pre-dose | 1.8 (7.69)
  SBP, Day 4 - Pre-dose | 1.8 (9.27)
  SBP, Day 5 | -2.9 (6.83)
  SBP, Day 6 | -3.9 (6.40)
  SBP, Day 7 | 0.3 (5.09)
  SBP, Day 8 | -4.4 (11.54)
  SBP, Follow-up | 1.5 (4.41)
  DBP, Day 2 - Pre-dose | -4.0 (5.45)
  DBP, Day 3 - Pre-dose | -0.3 (8.68)
  DBP, Day 4 - Pre-dose | -0.6 (8.86)
  DBP, Day 5 | -3.8 (8.66)
  DBP, Day 6 | -5.0 (7.84)
  DBP, Day 7 | -1.1 (7.62)
  DBP, Day 8 | -3.6 (4.50)
  DBP, Follow-up | 2.0 (7.46)

15. Primary Outcome: Change From Baseline in Vital Sign Parameters SBP and DBP for Part B
Description: Vital signs SBP and DBP were measured in the semi-supine position after 10 minutes of rest. Assessments were performed at Day 2 (pre-dose), Day 3 (pre-dose), Day 6, Day 9, Day 12, Day 15 and follow-up. Baseline was defined as assessments performed at Day 1(pre-dose). Change from Baseline was calculated as the post-dose visit value minus the Baseline value.
Time Frame: as for outcome 11
Population: Safety Population
Measure: Mean (Standard Deviation); unit: millimeters of mercury
Arm/Group | Part B-Placebo | Part B GSK2646264 1%
Number analyzed (Participants) | 3 | 9
millimeters of mercury
  SBP, Day 2 - Pre-dose | 8.3 (2.89) | 2.0 (6.60)
  SBP, Day 3 - Pre-dose | -1.7 (2.89) | 0.6 (8.82)
  SBP, Day 6 | 3.3 (2.89) | -1.3 (14.82)
  SBP, Day 9 | 5.0 (5.00) | -2.2 (10.64)
  SBP, Day 12 | 0.0 (0.00) | 1.4 (14.05)
  SBP, Day 15 | 8.3 (2.89) | -6.7 (11.73)
  SBP, Follow-up | 0.0 (0.00) | -3.3 (12.99)
  DBP, Day 2 - Pre-dose | 1.7 (10.41) | 2.4 (7.50)
  DBP, Day 3 - Pre-dose | 0.0 (8.66) | 0.8 (11.03)
  DBP, Day 6 | 0.0 (10.00) | 2.4 (14.05)
  DBP, Day 9 | -3.3 (7.64) | 3.6 (13.60)
  DBP, Day 12 | -3.3 (5.77) | 3.0 (9.60)
  DBP, Day 15 | -1.7 (11.55) | 2.4 (9.08)
  DBP, Follow-up | -1.7 (12.58) | 3.0 (13.77)

16. Primary Outcome: Change From Baseline in Vital Sign SBP and DBP for Part C
Description: Vital signs SBP and DBP were measured in the semi-supine position after 10 minutes of rest. Assessments were performed at Day 4 (pre-dose), Day 7 (pre-dose), Day 10, Day 15 and follow-up. Baseline was defined as assessments performed at Day 1 (pre-dose). Change from Baseline was calculated as the post-dose visit value minus the Baseline value. NA indicates standard deviation could not be calculated as a single participant was analyzed.
Time Frame: Baseline (Day 1 pre-dose) and Day 4 (pre-dose), Day 7 (pre-dose), Day 10, Day 15 and follow-up (Day 23)
Population: Safety Population
Measure: Mean (Standard Deviation); unit: millimeters of mercury
Arm/Group | Part C-Placebo | Part C GSK2646264 1%
Number analyzed (Participants) | 1 | 4
millimeters of mercury
  SBP, Day 4 - Pre-dose | -10.0 (NA) — NA indicates standard deviation could not be calculated as a single participant was analyzed. | -5.5 (12.56)
  SBP, Day 7 - Pre-dose | -10.0 (NA) — NA indicates standard deviation could not be calculated as a single participant was analyzed. | -4.5 (17.60)
  SBP, Day 10 | -10.0 (NA) — NA indicates standard deviation could not be calculated as a single participant was analyzed. | 5.3 (15.06)
  SBP, Day 15 | -10.0 (NA) — NA indicates standard deviation could not be calculated as a single participant was analyzed. | 12.3 (28.83)
  SBP, Follow-up | 0.0 (NA) — NA indicates standard deviation could not be calculated as a single participant was analyzed. | 10.0 (18.55)
  DBP, Day 4 - Pre-dose | -10.0 (NA) — NA indicates standard deviation could not be calculated as a single participant was analyzed. | -5.0 (9.13)
  DBP, Day 7 - Pre-dose | -10.0 (NA) — NA indicates standard deviation could not be calculated as a single participant was analyzed. | -4.8 (8.18)
  DBP, Day 10 | -20.0 (NA) — NA indicates standard deviation could not be calculated as a single participant was analyzed. | -6.5 (3.70)
  DBP, Day 15 | -10.0 (NA) — NA indicates standard deviation could not be calculated as a single participant was analyzed. | -1.0 (10.89)
  DBP, Follow-up | -10.0 (NA) — NA indicates standard deviation could not be calculated as a single participant was analyzed. | 2.0 (2.0)

17. Primary Outcome: Change From Baseline in Electrocardiogram (ECG) Parameters for Part A
Description: Triplicate 12-lead ECGs were obtained at screening and during the study single ECGs were taken. At each time point during the study ECG was taken using an ECG machine that automatically calculates the heart rate and measured the PR interval, QRS duration, corrected QT (QTc-Bazett [QTcB], QTC interval-Fredericia [QTcF]) intervals, RR interval and uncorrected QT interval. Baseline was defined as assessment performed at Day -1. Change from Baseline was calculated as the post-dose visit value minus the Baseline value.
Time Frame: Baseline (Day -1) and Day 4, and follow-up (Day 5 to Day 7)
Population: Safety Population
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Part A-GSK2646264 0.5%
Number analyzed (Participants) | 9
milliseconds
  PR interval, Day 4 | -0.67 (11.136)
  PR interval, Follow-up | 0.22 (12.347)
  QRS duration, Day 4 | -0.44 (5.637)
  QRS duration, Follow-up | -0.22 (5.239)
  QTcB, Day 4 | -6.11 (14.252)
  QTcB, Follow-up | -5.33 (16.963)
  QTcF, Day 4 | -1.22 (7.362)
  QTcF, Follow-up | -8.00 (13.829)
  RR interval, Day 4 | 82.89 (174.628)
  RR interval, Follow-up | -40.11 (114.704)
  Uncorrected QT Interval , Day 4 | 9.33 (23.302)
  Uncorrected QT Interval , Follow-up | -12.89 (20.028)

18. Primary Outcome: Change From Baseline in Electrocardiogram (ECG) Parameters for Part A
Description: Triplicate 12-lead ECGs were obtained at screening and during the study single ECGs were taken. At each time point during the study ECG was taken using an ECG machine that automatically calculates the heart rate and measured the PR interval, QRS duration, corrected QT (QTc-Bazett [QTcB], QTC interval-Fredericia[QTcF]) intervals, RR interval and uncorrected QT interval. Baseline was defined as assessment performed at Day -1. Change from Baseline was calculated as the post-dose visit value minus the Baseline value.
Time Frame: Baseline (Day -1) and Day 8 and follow-up (Day 9 to Day 11)
Population: Safety Population
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Part A-GSK2646264 1%
Number analyzed (Participants) | 8
milliseconds
  PR interval, Day 8 | 7.75 (17.678)
  PR interval, Follow-up | 4.00 (18.237)
  QRS duration, Day 8 | 0.25 (3.615)
  QRS duration, Follow-up | 3.25 (4.132)
  QTcB, Day 8 | -5.13 (10.696)
  QTcB, Follow-up | -1.75 (16.211)
  QTcF, Day 8 | -4.13 (8.855)
  QTcF, Follow-up | -5.63 (16.309)
  RR interval, Day 8 | 14.63 (88.569)
  RR interval, Follow-up | -49.75 (98.561)
  Uncorrected QT Interval , Day 8 | -2.00 (15.856)
  Uncorrected QT Interval , Follow-up | -13.00 (24.727)

19. Primary Outcome: Change From Baseline in ECG Parameters for Part B
Description: Triplicate 12-lead ECGs were obtained at screening and during the study single ECGs were taken. At each time point during the study ECG was taken using an ECG machine that automatically calculates the heart rate and measured the PR interval, QRS duration, QTcB, QTcF intervals, RR interval and uncorrected QT interval. Baseline was defined as assessment performed at Day -1. Change from Baseline was calculated as the post-dose visit value minus the Baseline value.
Time Frame: Baseline (Day -1) and Day 3 (pre-dose) and follow-up (Day 17 to Day 19)
Population: Safety Population
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Part B-Placebo | Part B GSK2646264 1%
Number analyzed (Participants) | 3 | 9
milliseconds
  PR interval, Day 3 Pre-dose | -6.67 (5.774) | 5.56 (10.138)
  PR interval, Follow-up | 3.33 (11.547) | -2.22 (10.929)
  QRS duration, Day 3 Pre-dose | -6.00 (12.166) | -2.44 (2.789)
  QRS duration, Follow-up | -4.67 (8.083) | -2.44 (3.127)
  QTcB, Day 3, Pre-dose | -13.00 (6.083) | -8.00 (17.428)
  QTcB, Follow-up | -5.33 (21.733) | -4.89 (11.185)
  QTcF, Day 3, Pre-dose | -6.33 (10.017) | -5.00 (11.203)
  QTcF, Follow-up | -3.00 (20.298) | -1.78 (6.906)
  RR interval, Day 3, Pre-dose | 95.33 (74.070) | 40.56 (131.342)
  RR interval, Follow-up | 30.00 (59.355) | 38.33 (86.510)
  Uncorrected QT Interval , Day 3, Pre-dose | 6.67 (19.218) | 0.67 (17.550)
  Uncorrected QT Interval , Follow-up | 1.33 (18.583) | 3.78 (10.745)

20. Primary Outcome: Change From Baseline in ECG Parameters for Part C
Description: Triplicate 12-lead ECGs were obtained at screening and during the study single ECGs were taken. At each time point during the study ECG was taken using an ECG machine that automatically calculates the heart rate and measured the PR interval, QRS duration, QTcB, QTcF intervals, RR interval and uncorrected QT interval. Baseline was defined as assessment performed at Day -1. Change from Baseline was calculated as the post-dose visit value minus the Baseline value. NA indicates standard deviation could not be calculated as a single participant was analyzed.
Time Frame: Baseline (Day -1) and Day 7 (pre-dose) and follow-up (Day 23)
Population: Safety Population
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Part C-Placebo | Part C GSK2646264 1%
Number analyzed (Participants) | 1 | 4
milliseconds
  PR interval, Day 7 Pre-dose | 10.00 (NA) — NA indicates standard deviation could not be calculated as a single participant was analyzed. | 1.50 (3.000)
  PR interval, Follow-up | -10.00 (NA) — NA indicates standard deviation could not be calculated as a single participant was analyzed. | -3.50 (4.726)
  QRS duration, Day 7 Pre-dose | -14.00 (NA) — NA indicates standard deviation could not be calculated as a single participant was analyzed. | -1.00 (1.155)
  QRS duration, Follow-up | -4.00 (NA) — NA indicates standard deviation could not be calculated as a single participant was analyzed. | 0.00 (1.633)
  QTcB, Day 7, Pre-dose | -14.00 (NA) — NA indicates standard deviation could not be calculated as a single participant was analyzed. | -4.50 (5.066)
  QTcB, Follow-up | -22.00 (NA) — NA indicates standard deviation could not be calculated as a single participant was analyzed. | 9.75 (17.557)
  QTcF, Day 7, Pre-dose | -6.00 (NA) — NA indicates standard deviation could not be calculated as a single participant was analyzed. | -3.25 (6.131)
  QTcF, Follow-up | -11.00 (NA) — NA indicates standard deviation could not be calculated as a single participant was analyzed. | 5.75 (12.920)
  RR interval, Day 7, Pre-dose | 115.00 (NA) — NA indicates standard deviation could not be calculated as a single participant was analyzed. | 17.50 (15.948)
  RR interval, Follow-up | 171.00 (NA) — NA indicates standard deviation could not be calculated as a single participant was analyzed. | -35.25 (117.766)
  Uncorrected QT Interval , Day 7, Pre-dose | 10.00 (NA) — NA indicates standard deviation could not be calculated as a single participant was analyzed. | -1.00 (7.394)
  Uncorrected QT Interval , Follow-up | 12.00 (NA) — NA indicates standard deviation could not be calculated as a single participant was analyzed. | -1.00 (16.452)

21. Primary Outcome: Number of Participants With Clinical Chemistry Data Outside the Range of Potential Clinical Importance (PCI) for Part A
Description: Clinical chemistry parameters assessed were alanine amino transferase (ALT), albumin (low <30 grams/liter), alkaline phosphatase, aspartate aminotransferase (AST), calcium (low <2 millimoles/liter and high >2.75 millimoles/liter), chloride, creatinine (high >159 micromoles/liter), direct bilirubin, gamma glutamyl transferase (GGT low <8 units/liter and high >78 units/liter), glucose (low <3 millimoles/liter and high >11.1 millimoles/liter), phosphorus (low 0.97 millimoles/liter and high 1.45 millimoles/liter), potassium (low <3 millimoles/liter and high >5.5 millimoles/liter), sodium (low <130 millimoles/liter and high >150 millimoles/liter), total bilirubin, total protein and urea/blood urea nitrogen (BUN). Values flagged as high and low of PCI for participants have been presented. Only categories with non-zero values have been presented.
Time Frame: Day 4 and follow up (Day 5 to Day 7)
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part A-GSK2646264 0.5%
Number analyzed (Participants) | 9
Participants | 1

22. Primary Outcome: Number of Participants With Clinical Chemistry Data Outside the Range of PCI for Part A
Description: Clinical chemistry parameters assessed were alanine amino transferase (ALT), albumin (low <30 grams/liter), alkaline phosphatase, AST, calcium (low <2 millimoles/liter and high >2.75 millimoles/liter), chloride, creatinine (high >159 micromoles/liter), direct bilirubin, GGT (low <8 units/liter and high >78 units/liter), glucose (low <3 millimoles/liter and high >11.1 millimoles/liter), phosphorus (low 0.97 millimoles/liter and high 1.45 millimoles/liter), potassium (low <3 millimoles/liter and high >5.5 millimoles/liter), sodium (low <130 millimoles/liter and high >150 millimoles/liter), total bilirubin, total protein and urea/BUN). Values flagged as high and low of PCI for participants have been presented. Only categories with non-zero values have been presented.
Time Frame: Day 5, Day 7 and follow up (Day 9 to Day 11)
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part A-GSK2646264 1%
Number analyzed (Participants) | 8
Participants
  Chloride, Day 5, High | 1
  Chloride, Day 7, High | 1
  Chloride, Follow-up, High, | 1
  GGT, Day 7, Low | 1

23. Primary Outcome: Number of Participants With Clinical Chemistry Data Outside the Range of PCI for Part B
Description: Clinical chemistry parameters assessed were ALT, albumin (low <30 grams/liter), alkaline phosphatase, AST, calcium (low <2 millimoles/liter and high >2.75 millimoles/liter), chloride (low <98 millimoles/liter and high >106 millimoles/liter), creatinine (high >159 micromoles/liter), direct bilirubin, GGT (low <8 units/liter and high >78 units/liter), glucose (low <3 millimoles/liter and high >11.1 millimoles/liter), phosphorus (low 0.97 millimoles/liter and high 1.45 millimoles/liter), potassium (low <3 millimoles/liter and high >5.5 millimoles/liter), sodium (low <130 millimoles/liter and high >150 millimoles/liter), total bilirubin, total protein and urea/BUN (low <2.9 and high >7.1). Values flagged as high and low of PCI for participants have been presented. Only categories with non-zero values have been presented.
Time Frame: Day 3 and follow up (Day 17 to Day 19)
Population: Safety Population. Only those participants with data available at the specified time points were analyzed (represented by n=x in the category titles).
Measure: Count of Participants; unit: Participants
Arm/Group | Part B-Placebo | Part B GSK2646264 1%
Number analyzed (Participants) | 3 | 9
Participants
  Chloride, Day 3, Low, n=3,9 | 1 | 1
  Chloride, Follow up, Low,n=3,9 | 3 | 1
  Chloride, Follow-up, High, n=3,9 | 0 | 1
  Direct Bilirubin, Day 3, High, n=3,8: number analyzed (Participants) | 3 | 8
  Direct Bilirubin, Day 3, High, n=3,8 | 0 | 1
  Direct Bilirubin, Follow-up, High, n=3,9 | 0 | 1
  GGT, Day 3, High, n=3,9 | 0 | 1
  GGT, Follow-up, Low, n=3,9 | 1 | 0
  Phosphorus, Day 3, Low, n=3,9 | 1 | 4
  Phosphorus, Follow-up, Low, n=3,9 | 1 | 3
  Potassium, Day 3, Low, n=3,9 | 0 | 1
  Potassium, Day 3, High, n=3,9 | 1 | 0
  Potassium, Follow-up, Low, n=3,9 | 0 | 1
  Urea/BUN, Day 3, Low, n=3,9 | 0 | 1
  Urea/BUN, Follow-up, High, n=3,8: number analyzed (Participants) | 3 | 8
  Urea/BUN, Follow-up, High, n=3,8 | 1 | 0

24. Primary Outcome: Number of Participants With Clinical Chemistry Data Outside the Range of PCI for Part C
Description: Clinical chemistry parameters assessed were ALT, albumin (low <30 grams/liter), alkaline phosphatase, AST, calcium (low <2 millimoles/liter and high >2.75 millimoles/liter), chloride (low <98 millimoles/liter and high >106 millimoles/liter), creatinine (high >159 micromoles/liter), direct bilirubin, GGT (low <8 units/liter and high >78 units/liter), glucose (low <3 millimoles/liter and high >11.1 millimoles/liter), phosphorus (low 0.97 millimoles/liter and high 1.45 millimoles/liter), potassium (low <3 millimoles/liter and high >5.5 millimoles/liter), sodium (low <130 millimoles/liter and high >150 millimoles/liter), total bilirubin, total protein (low <60 grams/liter and high >78 grams/liter) and urea/BUN (low <2.9 millimoles/liter and high >7.1 millimoles/liter). Values flagged as high and low of PCI for participants have been presented. Only categories with non-zero values have been presented.
Time Frame: Day 1, Day 7 and follow up (Day 23)
Population: as for outcome 23
Measure: Count of Participants; unit: Participants
Arm/Group | Part C-Placebo | Part C GSK2646264 1%
Number analyzed (Participants) | 1 | 4
Participants
  Chloride, Day 7, Low, n=1,2: number analyzed (Participants) | 1 | 2
  Chloride, Day 7, Low, n=1,2 | 1 | 0
  Chloride, Follow-up, Low, n=1,3: number analyzed (Participants) | 1 | 3
  Chloride, Follow-up, Low, n=1,3 | 0 | 1
  Phosphorus, Day 1, Low, n=1,4 | 0 | 1
  Urea/BUN, Day 1, Low, n=1,2: number analyzed (Participants) | 1 | 2
  Urea/BUN, Day 1, Low, n=1,2 | 0 | 1
  Total protein, Day 1, High, n=1,4 | 0 | 1

25. Primary Outcome: Number of Participants With Hematology Data Outside the Range of PCI for Part A
Description: Hematology parameters assessed were basophils (high >0.1x10^9 cells/Liter), eosinophils (high >0.44x 10^9 cells/Liter), hematocrit, hemoglobin, lymphocytes (low <0.8x10^9 cells/Liter), mean corpuscle hemoglobin (MCH low <28 picograms and high >32 picograms), mean corpuscle hemoglobin concentration (MCHC low <32 grams/liter and high >36 grams/liter), mean corpuscle volume (MCV), monocytes (high >0.208x 10^9 cells/Liter), platelet count, red blood cell (RBC low <4.2x10^6 cells/microliter and high 5.9x10^6 cells/microliter) count, total neutrophils and white blood cell (WBC) count. Values flagged as high and low of PCI for participants have been presented. Only categories with non-zero values have been presented.
Time Frame: Day 4 and follow up (Day 5 to Day 7)
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part A-GSK2646264 0.5%
Number analyzed (Participants) | 9
Participants
  Basophils, Day 4, High | 9
  Basophils, Follow-up, High | 9
  Eosinophils, Day 4, High | 1
  MCH, Day 4, High | 1
  MCH, Follow-up, High | 1
  Monocytes, Day 4, High | 9
  Monocytes, Follow-up, High | 9
  Lymphocytes, Follow-up, Low | 0
  RBC count, Follow-up, Low | 0

26. Primary Outcome: Number of Participants With Hematology Data Outside the Range of PCI for Part A
Description: Hematology parameters assessed were basophils (high >0.1x10^9 cells/Liter), eosinophils (high >0.44x 10^9 cells/Liter), hematocrit, hemoglobin, lymphocytes (low <0.8x10^9 cells/Liter), MCH (low <28 picograms and high >32 picograms), MCHC (low <32 grams/liter and high >36 grams/liter), MCV, monocytes (high >0.208x10^9 cells/Liter), platelet count, RBC count (low <4.2x10^6 cells/microliter and high 5.9x10^6 cells/microliter) count, total neutrophils, WBC count. Values flagged as high and low of PCI for participants have been presented. Only categories with non-zero values have been presented.
Time Frame: Day 5, Day 7 and follow up (Day 9 to Day 11)
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part A-GSK2646264 1%
Number analyzed (Participants) | 8
Participants
  Basophils, Day 5, High | 7
  Basophils, Day 7, High | 8
  Basophils, Follow-up, High | 8
  MCH, Follow-up, High | 0
  MCHC, Day 5, High | 1
  MCHC, Day 7, High | 1
  Monocytes, Day 5, High | 8
  Monocytes, Day 7, High | 8
  Monocytes, Follow-up, High | 8
  Lymphocytes, Follow-up,Low | 1
  RBC count, Day 5, Low | 1
  RBC count, Day 7, Low | 1
  RBC count, Follow-up, Low | 1

27. Primary Outcome: Number of Participants With Hematology Data Outside the Range of PCI for Part B
Description: Hematology parameters assessed were basophils (high >0.1x10^9 cells/Liter), eosinophils (high >0.44x 10^9 cells/Liter), hematocrit, hemoglobin, lymphocytes (low <0.8x10^9 cells/Liter), MCH (low <28 picograms and high >32 picograms), MCHC (low <32 grams/liter and high >36 grams/liter), MCV, monocytes (high >0.208x10^9 cells/Liter), platelet count, RBC count (low <4.2x10^6 cells/microliter and high 5.9x10^6 cells/microliter) count, total neutrophils and WBC count. Values flagged as high and low of PCI for participants have been presented. Only categories with non-zero values have been presented.
Time Frame: Day 3 and follow up (Day 17 to 19)
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part B-Placebo | Part B GSK2646264 1%
Number analyzed (Participants) | 3 | 9
Participants
  Basophils, Day 3, High | 3 | 9
  Basophils, Follow-up, High | 3 | 9
  Eosinophils, Day 3, High | 0 | 1
  Eosinophils, Follow-up, High | 0 | 1
  Monocytes, Day 3, High | 3 | 9
  Monocytes, Follow-up, High | 3 | 9
  MCHC, Follow-up, Low | 0 | 1
  RBC count, Follow-up, Low | 1 | 0

28. Primary Outcome: Number of Participants With Hematology Data Outside the Range of PCI for Part C
Description: Hematology parameters assessed were basophils (high >0.1x10^9 cells/Liter), eosinophils (high >0.44x 10^9 cells/Liter), hematocrit, hemoglobin, lymphocytes (low <0.8x10^9 cells/Liter), MCH (low <28 picograms and high >32 picograms), MCHC low <32 grams/liter and high >36 grams/liter), MCV, monocytes (high >0.208x10^9 cells/Liter), platelet count, RBC count (low <4.2x10^6 cells/microliter and high 5.9x10^6 cells/microliter) count, total neutrophils and WBC count. Values flagged as high and low of PCI for participants have been presented. Only categories with non-zero values have been presented.
Time Frame: Day 1, Day 7 and follow up (Day 23)
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part C-Placebo | Part C GSK2646264 1%
Number analyzed (Participants) | 1 | 4
Participants
  Basophils, Day 1, High | 1 | 3
  Basophils, Day 7, High | 1 | 3
  Basophils, Follow-up, High | 1 | 2
  Monocytes, Day 1, High | 1 | 4
  Monocytes, Day 7, High | 1 | 4
  Monocytes, Follow-up, High | 1 | 4
  MCH, Day 1, Low | 1 | 0
  MCH, Day 7, Low | 1 | 0
  MCH, Follow-up, Low | 1 | 0

29. Primary Outcome: Number of Participants With Tolerability Assessment for Part A
Description: Tolerability was assessed with the skin irritation scoring system of study, where the score consists of a numeric score according to the dermal response scoring as follows 0=no evidence of irritation, 1=minimal erythema, barely perceptible (pink), 2=moderate erythema (definite redness), 3=strong erythema (intense redness), 4=definite edema, 5=erythema, edema, and papules, 6=vesicular eruption, 7=strong reaction spreading beyond test site, and a letter according to the other effects scoring, Z=no other effect, A=slight glazed appearance, B=marked glazing, C=glazing with peeling and cracking, F=glazing with fissures, G=film of dried serous exudate covering all or part of the patch site, H=small petechial erosions and/or scabs. For each skin assessment, letter grade will be converted to numeric values as below: A=0, Z=0, B=1, C=2, F=3, G=3, H=3. A combined score for each participant was calculated by adding all numeric and letter scores. A maximum score of 3 was allowed.
Time Frame: Up to Day 4
Population: Safety Population
Measure: Count of Participants; unit: Participants
Groups:
- Part A-Placebo (Group 1): Participants were treated topically with matching placebo cream on an area of approximately 12 x 3 cm on the volar aspect of the arm which approximated to 0.2% total BSA, on each arm. On Day 2 and Day 3 participants received active treatment and placebo on the same arms as on Day 1, with the percentage BSA being 1% on Day 2 and 5% on Day 3.
- Part A-GSK2646264 0.5% (Group 1): Participants were treated topically with GSK2646264 0.5% cream on an area of approximately 12 x 3 cm on the volar aspect of the arm which approximated to 0.2% total BSA, on each arm. On Day 2 and Day 3 participants received active treatment and placebo on the same arms as on Day 1, with the percentage BSA being 1% on Day 2 and 5% on Day 3.
- Part A-Placebo (Group 2): Participants received placebo on Days 1, 2, 3 and 4. On Day 1 and Day 2, participants received treatment to 0.2% BSA; placebo treatment to one arm. In addition, participants received treatment to another 5% BSA; placebo to one side of the torso. On Days 3 and 4, the same treatment to the arms was applied as on Days 1 and 2, but the %BSA of the torso to which treatment was applied to was increased to 10%.
- Part A-GSK2646264 1% (Group 2): Participants received active treatment (1% cream strength) on Days 1, 2, 3 and 4. On Day 1 and Day 2, participants received treatment to 0.2% BSA; active treatment on one arm. In addition, participants received treatment to another 5% BSA; active to one side of the torso. On Days 3 and 4, the same treatment to the arms was applied as on Days 1 and 2, but the %BSA of the torso to which treatment was applied to was increased to 10%.
Arm/Group | Part A-Placebo (Group 1) | Part A-GSK2646264 0.5% (Group 1) | Part A-Placebo (Group 2) | Part A-GSK2646264 1% (Group 2)
Number analyzed (Participants) | 9 | 9 | 8 | 8
Participants
  Maximal dermal response, Grade 0 | 9 | 8 | 6 | 8
  Maximal dermal response, Grade 1 | 0 | 1 | 2 | 0
  Maximal dermal response, Grade 2 | 0 | 0 | 0 | 0
  Maximal dermal response, Grade 3 | 0 | 0 | 0 | 0
  Maximal dermal response, Grade 4 | 0 | 0 | 0 | 0
  Maximal dermal response, Grade 5 | 0 | 0 | 0 | 0
  Maximal dermal response, Grade 6 | 0 | 0 | 0 | 0
  Maximal dermal response, Grade 7 | 0 | 0 | 0 | 0
  Maximal other dermal effects, Z | 9 | 9 | 8 | 8
  Maximal other dermal effects, A | 0 | 0 | 0 | 0
  Maximal other dermal effects, B | 0 | 0 | 0 | 0
  Maximal other dermal effects, C | 0 | 0 | 0 | 0
  Maximal other dermal effects, F | 0 | 0 | 0 | 0
  Maximal other dermal effects, G | 0 | 0 | 0 | 0
  Maximal other dermal effects, H | 0 | 0 | 0 | 0

30. Primary Outcome: Number of Participants With Tolerability Assessment for Part B
Description: as for outcome 29
Time Frame: Up to Day 3
Measure: Count of Participants; unit: Participants
Arm/Group | Part B (10% BSA)-Placebo | Part B (10% BSA) GSK2646264 1% | Part B (3.5% BSA)-Placebo | Part B (3.5% BSA) GSK2646264 1%
Number analyzed (Participants) | 1 | 3 | 2 | 6
Participants
  Maximal dermal response, Grade 0 | 0 | 0 | 2 | 6
  Maximal dermal response, Grade 1 | 0 | 1 | 0 | 0
  Maximal dermal response, Grade 2 | 1 | 0 | 0 | 0
  Maximal dermal response, Grade 3 | 0 | 1 | 0 | 0
  Maximal dermal response, Grade 4 | 0 | 1 | 0 | 0
  Maximal dermal response, Grade 5 | 0 | 0 | 0 | 0
  Maximal dermal response, Grade 6 | 0 | 0 | 0 | 0
  Maximal dermal response, Grade 7 | 0 | 0 | 0 | 0
  Maximal other dermal effects, Z | 1 | 2 | 2 | 6
  Maximal other dermal effects, A | 0 | 0 | 0 | 0
  Maximal other dermal effects, B | 0 | 1 | 0 | 0
  Maximal other dermal effects, C | 0 | 0 | 0 | 0
  Maximal other dermal effects, F | 0 | 0 | 0 | 0
  Maximal other dermal effects, G | 0 | 0 | 0 | 0
  Maximal other dermal effects, H | 0 | 0 | 0 | 0

31. Primary Outcome: Number of Participants With Tolerability Assessment for Part C
Description: as for outcome 29
Time Frame: Up to Day 7
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Part C-Placebo | Part C GSK2646264 1%
Number analyzed (Participants) | 1 | 4
Participants
  Maximal dermal response, Grade 0 | 1 | 4
  Maximal dermal response, Grade 1 | 0 | 0
  Maximal dermal response, Grade 2 | 0 | 0
  Maximal dermal response, Grade 3 | 0 | 0
  Maximal dermal response, Grade 4 | 0 | 0
  Maximal dermal response, Grade 5 | 0 | 0
  Maximal dermal response, Grade 6 | 0 | 0
  Maximal dermal response, Grade 7 | 0 | 0
  Maximal other dermal effects, Z | 1 | 4
  Maximal other dermal effects, A | 0 | 0
  Maximal other dermal effects, B | 0 | 0
  Maximal other dermal effects, C | 0 | 0
  Maximal other dermal effects, F | 0 | 0
  Maximal other dermal effects, G | 0 | 0
  Maximal other dermal effects, H | 0 | 0

32. Secondary Outcome: Plasma GSK2646264 Pharmacokinetic (PK) Concentrations for Part A
Description: Blood samples were collected to assess the plasma concentration of GSK2646264 for Part A on Day 1 (Pre-dose,1,2,4,8,12,24 hours), Day 2 (1,2,4,8,12,24 hours) and Day 3 (1,2,4,8,12,24 hours). The actual date and time of each blood sample collection was recorded. PK Population comprised of all randomized participants of the Safety Population for whom a pharmacokinetic sample was obtained and analyzed.
Time Frame: Day 1 (Pre-dose,1,2,4,8,12,24 hours), Day 2 (1,2,4,8,12,24 hours) and Day 3 (1,2,4,8,12,24 hours)
Population: PK Population
Measure: Mean (Standard Deviation); unit: nanograms/milliliter
Arm/Group | Part A-GSK2646264 0.5%
Number analyzed (Participants) | 9
nanograms/milliliter
  Day 1, Pre-dose | 0.00000 (0.00000)
  Day 1, 1 hour | 0.00000 (0.00000)
  Day 1, 2 hours | 0.00000 (0.00000)
  Day 1, 4 hours | 0.00000 (0.00000)
  Day 1, 8 hours | 0.00000 (0.00000)
  Day 1, 12 hours | 0.00708 (0.021233)
  Day 1, 24 hours | 0.02457 (0.039577)
  Day 2, 1 hour | 0.00600 (0.018000)
  Day 2, 2 hours | 0.02524 (0.038068)
  Day 2, 4 hours | 0.07198 (0.064932)
  Day 2, 8 hours | 0.20567 (0.340281)
  Day 2, 12 hours | 0.16524 (0.117680)
  Day 2, 24 hours | 0.23991 (0.092812)
  Day 3, 1 hour | 0.25198 (0.105292)
  Day 3, 2 hours | 0.36364 (0.197974)
  Day 3, 4 hours | 0.50156 (0.239403)
  Day 3, 8 hours | 0.67546 (0.396632)
  Day 3, 12 hours | 0.81486 (0.463918)
  Day 3, 24 hours | 1.03606 (0.601077)

33. Secondary Outcome: Plasma GSK2646264 Pharmacokinetic (PK) Concentrations for Part A
Description: Blood samples were collected to assess the plasma concentration of GSK2646264 for Part A on Day 1 (Pre-dose,1,2,4,8,12,24 hours), Day 2 (1,2,4,8,12,24 hours), Day 3 (1,2,4,8,12,24 hours) and Day 4 post-dose at Day 5 (30 and 36 hours), Day 6 (48,54 and 60 hours), Day 7 (72,78 and 84 hours) and Day 8 (96 hours). The actual date and time of each blood sample collection was recorded.
Time Frame: Day 1 (Pre-dose,1,2,4,8,12,24 hours), Day 2 (1,2,4,8,12,24 hours), Day 3 (1,2,4,8,12,24 hours) and Day 4 post-dose at Day 5 (30 and 36 hours), Day 6 (48,54 and 60 hours), Day 7 (72,78 and 84 hours) and Day 8 (96 hours)
Measure: Mean (Standard Deviation); unit: nanograms/milliliter
Groups:
- Part A-GSK2646264 1%: Participants were treated topically with 0.5 % GSK2646264 cream and placebo cream on an area of approximately 12 x 3 cm on the volar aspect of the arm which approximated to 0.2% total BSA, on each arm. On Day 2 and Day 3 participants received active treatment and placebo on the same arms as on Day 1, with the percentage BSA being 1% on Day 2 and 5% on Day 3.
Arm/Group | Part A-GSK2646264 1%
Number analyzed (Participants) | 8
nanograms/milliliter
  Day 1, Pre-dose | 0.00000 (0.00000)
  Day 1, 1 hour | 0.00000 (0.00000)
  Day 1, 2 hours | 0.02780 (0.02780)
  Day 1, 4 hours | 0.19470 (0.19470)
  Day 1, 8 hours | 0.31849 (0.31849)
  Day 1, 12 hours | 0.49735 (0.49735)
  Day 1, 24 hours | 0.86538 (0.86538)
  Day 2, 1 hour | 0.82164 (0.82164)
  Day 2, 2 hours | 0.91896 (0.91896)
  Day 2, 4 hours | 1.10081 (1.10081)
  Day 2, 8 hours | 1.18935 (1.18935)
  Day 2, 12 hours | 1.44756 (1.44756)
  Day 2, 24 hours | 2.11824 (2.11824)
  Day 3, 1 hour | 2.15994 (2.15994)
  Day 3, 2 hours | 2.17775 (2.17775)
  Day 3, 4 hours | 2.39909 (2.39909)
  Day 3, 8 hours | 2.30511 (2.30511)
  Day 3, 12 hours | 2.72968 (2.72968)
  Day 3, 24 hours | 3.40905 (3.40905)
  Day 4, 1 hour | 3.64494 (3.64494)
  Day 4, 2 hours | 3.76981 (3.76981)
  Day 4, 4 hours | 3.99425 (3.99425)
  Day 4, 8 hours | 3.88128 (3.88128)
  Day 4, 12 hours | 4.13984 (4.13984)
  Day 4, 24 hours | 5.35715 (5.35715)
  Day 5, 30 hours | 4.98988 (1.807766)
  Day 5, 36 hours | 4.63755 (1.629070)
  Day 6, 48 hours | 4.92234 (1.690833)
  Day 6, 54 hours | 4.44403 (1.834524)
  Day 6, 60 hours | 4.04828 (1.646939)
  Day 7, 72 hours | 4.02665 (1.592538)
  Day 7, 78 hours | 3.76244 (1.751219)
  Day 7, 84 hours | 3.45551 (1.522890)
  Day 8, 96 hours | 3.30003 (1.364104)

34. Secondary Outcome: Plasma GSK2646264 PK Concentrations for Part B
Description: Blood samples were collected to assess the plasma concentration of GSK2646264 for Part B on Day 1 (Pre-dose,1,4,8,12,24 hours), Day 2 (1,4,8,12,24 hours), Day 3 (1,4,8,12,24 hours), Day 6, Day 9, Day 12, Day 15 and follow-up (Day 17 to 19). The actual date and time of each blood sample collection was recorded.
Time Frame: Day 1 (Pre-dose,1,4,8,12,24 hours), Day 2 (1,4,8,12,24 hours), Day 3 (1,4,8,12,24 hours), Day 6, Day 9, Day 12, Day 15 and follow-up (Day 17 to 19)
Population: PK Population
Measure: Mean (Standard Deviation); unit: nanograms/milliliter
Groups:
- Part B (10% BSA) GSK2646264 1%: CU participants received matching placebo treatment to an area of 10% BSA (5% BSA each arm) on Days 1, 2 and 3.
Arm/Group | Part B (10% BSA) GSK2646264 1% | Part B (3.5% BSA) GSK2646264 1%
Number analyzed (Participants) | 3 | 6
nanograms/milliliter
  Day 1, Pre-dose | 0.00000 (0.00000) | 0.00000 (0.00000)
  Day 1, 1 hour | 0.00000 (0.00000) | 0.01083 (0.026536)
  Day 1, 4 hours | 0.61280 (0.640458) | 0.21290 (0.236751)
  Day 1, 8 hours | 2.22747 (1.658949) | 0.67952 (0.529431)
  Day 1, 12 hours | 2.72833 (2.378997) | 1.51255 (1.018452)
  Day 1, 24 hours | 3.06623 (1.944608) | 1.44370 (0.845724)
  Day 2, 1 hour | 3.02890 (1.739913) | 1.63247 (0.903514)
  Day 2, 4 hours | 3.63953 (1.603219) | 1.86712 (0.891829)
  Day 2, 8 hours | 4.01943 (1.338776) | 2.28577 (1.202992)
  Day 2, 12 hours | 4.76710 (0.642243) | 2.57673 (1.451027)
  Day 2, 24 hours | 5.04110 (0.124156) | 2.90163 (1.598613)
  Day 3, 1 hour | 5.15953 (0.564893) | 3.09353 (1.715172)
  Day 3, 4 hours | 6.38943 (1.585360) | 3.38355 (1.765959)
  Day 3, 8 hours | 6.35937 (1.256342) | 3.30380 (1.694633)
  Day 3, 12 hours | 6.73903 (1.011669) | 3.60315 (2.004840)
  Day 3, 24 hours | 8.84147 (1.665464) | 4.29153 (2.451293)
  Day 6 | 3.54063 (0.611174) | 2.14953 (1.053739)
  Day 9 | 1.89157 (0.453369) | 1.00005 (0.572714)
  Day 12 | 0.82347 (0.545903) | 0.57632 (0.320586)
  Day 15 | 0.42230 (0.195058) | 0.28658 (0.232548)
  Follow-up | 0.22513 (0.129284) | 0.12982 (0.105350)

35. Secondary Outcome: Plasma GSK2646264 PK Concentrations for Part C
Description: Blood samples were collected to assess the plasma concentration of GSK2646264 for Part C on Day 1 (Pre-dose,1 and 4 hours), Day 4 (Pre-dose and 4 hours), Day 7 (Pre-dose and 4 hours), Day 10, Day 15 and follow-up. The actual date and time of each blood sample collection was recorded.
Time Frame: Day 1 (Pre-dose,1 and 4 hours), Day 4 (Pre-dose and 4 hours), Day 7 (Pre-dose and 4 hours), Day 10, Day 15 and follow-up (Day 23)
Population: PK Population. Only those participants with data available at the specified time points were analyzed (represented by n=x in the category titles).
Measure: Mean (Standard Deviation); unit: nanograms/milliliter
Arm/Group | Part C GSK2646264 1%
Number analyzed (Participants) | 4
nanograms/milliliter
  Day 1, Pre-dose, n=3: number analyzed (Participants) | 3
  Day 1, Pre-dose, n=3 | 0.00000 (0.00000)
  Day 1, 4 hours, n=4 | 0.18048 (0.123670)
  Day 4, Pre-dose, n=3: number analyzed (Participants) | 3
  Day 4, Pre-dose, n=3 | 1.22397 (0.963854)
  Day 4, 4 hours, n=3: number analyzed (Participants) | 3
  Day 4, 4 hours, n=3 | 1.37440 (0.961820)
  Day 7, Pre-dose, n=4 | 2.33635 (2.342202)
  Day 7, 4 hours, n=4 | 2.77940 (2.275138)
  Day 10,n=4 | 2.13075 (1.830816)
  Day 15,n=4 | 0.91718 (0.895466)
  Follow-up, n=4 | 0.44233 (0.349810)

36. Secondary Outcome: Area Under the Concentration-time Curve From Time 0 to t (AUC [0-t]) of GSK2646264 for Part A
Description: Blood samples were collected at the indicated time point to investigate the PK profile of GSK264624. From the GSK2646264 concentration-time data, the AUC (0-T) was determined using the currently approved and validated software.
Time Frame: Pre dose, 1 ,2, 4, 8, 12 and 24 hours post-dose on Days 1,2 and Day 3
Population: PK Population. Only those participants with data available at the specified time points were analyzed represented by n=x in the category titles).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanograms/milliliter
Groups:
- Part A-GSK2646264 0.5%: Participants were treated topically with GSK2646264 0.5% cream on an area of approximately 12 x 3 cm on the volar aspect of the arm which approximated to 0.2% total BSA, on each arm. On Day 2 and Day 3 participants recieved active treatment and placebo on the same arms as on Day 1, with the percentage BSA being 1% on Day 2 and 5% on Day 3.
Arm/Group | Part A-GSK2646264 0.5%
Number analyzed (Participants) | 9
Hours*nanograms/milliliter
  Day 1, n=3: number analyzed (Participants) | 3
  Day 1, n=3 | 0.5411 (45)
  Day 2,n=9 | 3.1462 (60)
  Day 3, n=9 | 15.2614 (66)

37. Secondary Outcome: AUC (0-t) of GSK2646264 for Part A
Description: as for outcome 36
Time Frame: Day 1 (Pre-dose,1,2,4,8,12,24 hours), Day 2 (Pre-dose,1,2,4,8,12,24 hours), Day 3 (Pre-dose,1,2,4,8,12,24 hours) and Day 4 post-dose
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanograms/milliliter
Arm/Group | Part A-GSK2646264 1%
Number analyzed (Participants) | 8
Hours*nanograms/milliliter
  Day 1 | 8.6870 (86)
  Day 2 | 31.0600 (53)
  Day 3 | 60.2293 (40)
  Day 4 | 382.4520 (40)

38. Secondary Outcome: Maximum Plasma Concentration (Cmax) of GSK2646264 for Part A
Description: Blood samples were collected at the indicated time point to investigate the PK profile of GSK264624. From the GSK2646264 concentration-time data, the Cmax was determined using the currently approved and validated software.
Time Frame: Pre dose, 1 ,2, 4, 8, 12 and 24 hours post-dose on Days 1,2 and Day 3
Population: as for outcome 36
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms/milliliter
Arm/Group | Part A-GSK2646264 0.5%
Number analyzed (Participants) | 9
Nanograms/milliliter
  Day 1, n=3: number analyzed (Participants) | 3
  Day 1, n=3 | 0.07360 (34)
  Day 2, n=9 | 0.25084 (69)
  Day 3,n=9 | 0.90382 (69)

39. Secondary Outcome: Cmax of GSK2646264 for Part A
Description: Blood samples were collected at the indicated time points to investigate the PK profile of GSK264624. From the GSK2646264 concentration-time data, the Cmax was determined using the currently approved and validated software.
Time Frame: as for outcome 37
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms/milliliter
Arm/Group | Part A-GSK2646264 1%
Number analyzed (Participants) | 8
Nanograms/milliliter
  Day 1 | 0.72391 (72)
  Day 2 | 1.96715 (43)
  Day 3 | 3.28320 (34)
  Day 4 | 5.22144 (41)

40. Secondary Outcome: Area Under the Concentration-time Curve From Time 0 to 24 Hours (AUC [0-24]) of GSK2646264 for Part A
Description: Blood samples were collected at the indicated time point to investigate the PK profile of GSK264624. From the GSK2646264 concentration-time data, the AUC (0-24) was determined using the currently approved and validated software. NA indicated data was not collected due to insufficient participants with data.
Time Frame: Pre dose, 1 ,2, 4, 8, 12 and 24 hours post-dose on Days 1,2,3 and 4
Population: PK Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanograms/milliliter
Arm/Group | Part A-GSK2646264 0.5%
Number analyzed (Participants) | 9
Hours*nanograms/milliliter | NA (NA) — NA indicated data was not collected due to insufficient participants with data.

41. Secondary Outcome: Area Under the Concentration-time Curve From Time 0 to 24 Hours (AUC [0-24]) of GSK2646264 for Part A
Description: Blood samples were collected at the indicated time point to investigate the PK profile of GSK264624. From the GSK2646264 concentration-time data, the AUC (0-24) was determined using the currently approved and validated software.
Time Frame: Pre dose, 1 ,2, 4, 8, 12 and 24 hours post-dose on Days 1,2,3 and 4
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanograms/milliliter
Arm/Group | Part A-GSK2646264 1%
Number analyzed (Participants) | 8
Hours*nanograms/milliliter | 97.8835 (37)

42. Secondary Outcome: Time to Cmax (Tmax) of GSK2646264 for Part A
Description: Blood samples were collected at the indicated time points to investigate the PK profile of GSK264624. From the GSK2646264 concentration-time data, the tmax was determined using the currently approved and validated software.
Time Frame: Pre dose, 1 ,2, 4, 8, 12 and 24 hours post-dose on Days 1,2 and Day 3
Population: as for outcome 36
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Part A-GSK2646264 0.5%
Number analyzed (Participants) | 9
hours
  Day 1, n=3: number analyzed (Participants) | 3
  Day 1, n=3 | 19.60 (6.585)
  Day 2, n=9 | 21.52 (5.074)
  Day 3,n=9 | 20.32 (7.267)

43. Secondary Outcome: Tmax of GSK2646264 for Part A
Description: Blood samples were collected at the indicated time point to investigate the PK profile of GSK264624. From the GSK2646264 concentration-time data, the tmax was determined using the currently approved and validated software.
Time Frame: as for outcome 37
Population: PK Population
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Part A-GSK2646264 1%
Number analyzed (Participants) | 8
hours
  Day 1 | 23.85 (0.053)
  Day 2 | 23.83 (0.046)
  Day 3 | 22.29 (4.158)
  Day 4 | 28.99 (14.180)

44. Secondary Outcome: Terminal Half-life (t1/2) of GSK2646264 for Part A
Description: Blood samples were collected at the indicated time point to investigate the PK profile of GSK264624. From the GSK2646264 concentration-time data, the t1/2 was determined using the currently approved and validated software. NA indicated t1/2 could not be calculated as we need at least 3 time points after Cmax within the same participant and this criteria could not be fulfilled due to lack of available data.
Time Frame: Pre dose, 1 ,2, 4, 8, 12 and 24 hours post-dose on Days 1,2,3 and 4
Population: PK Population
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Part A-GSK2646264 0.5%
Number analyzed (Participants) | 9
hours | NA (NA) — NA indicated t1/2 could not be calculated as we need at least 3 time points after Cmax within the same participant and this criteria could not be fulfilled due to lack of available data.

45. Secondary Outcome: t1/2 of GSK2646264 for Part A
Description: as for outcome 44
Time Frame: Day 1 (Pre-dose,1,2,4,8,12,24 hours), Day 2 (Pre-dose,1,2,4,8,12,24 hours), Day 3 (Pre-dose,1,2,4,8,12,24 hours) and Day 4 post-dose at Day 5 (30 and 36 hours), Day 6 (48,54 and 60 hours), Day 7 (72,78 and 84 hours) and Day 8 (96 hours)
Population: PK Population
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Part A-GSK2646264 1%
Number analyzed (Participants) | 8
hours | NA (NA) — NA indicated t1/2 could not be calculated as we need at least 3 time points after Cmax within the same participant and this criteria could not be fulfilled due to lack of available data.

46. Secondary Outcome: AUC [0-t] of GSK2646264 for Part B
Description: as for outcome 36
Time Frame: Pre dose, 1 ,2, 4, 8, 12 hours post-dose on Days 1,2,3 and 24 hours post last dose on Day 3
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanograms/milliliter
Arm/Group | Part B (10% BSA) GSK2646264 1% | Part B (3.5% BSA) GSK2646264 1%
Number analyzed (Participants) | 3 | 6
Hours*nanograms/milliliter
  Day 1 | 40.5235 (92) | 18.7840 (101)
  Day 2 | 100.6152 (18) | 46.5654 (96)
  Day 3 | 825.1809 (22) | 379.8602 (109)

47. Secondary Outcome: Cmax of GSK2646264 for Part B
Description: as for outcome 38
Time Frame: Pre dose, 1 ,2, 4, 8, 12 hours post-dose on Days 1,2,3 and 24 hours post last dose on Day 3 (Day 4)
Population: PK Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms/milliliter
Arm/Group | Part B (10% BSA) GSK2646264 1% | Part B (3.5% BSA) GSK2646264 1%
Number analyzed (Participants) | 3 | 6
Nanograms/milliliter
  Day 1 | 2.71563 (69) | 1.30673 (109)
  Day 2 | 5.14144 (6) | 2.41207 (92)
  Day 3 | 7.51684 (8) | 2.89771 (120)

48. Secondary Outcome: AUC (0-24) of GSK2646264 for Part B
Description: Blood samples were collected at the indicated time point to investigate the PK profile of GSK264624. From the GSK2646264 concentration-time data, the AUC (0-24) was determined using the currently approved and validated software. NA indicates that geometric coefficient of variation could not be computed for Part B (3.5% BSA) GSK2646264 1% as a single participant was analyzed on Day 2.
Time Frame: Pre dose, 1 ,2, 4, 8, 12 hours post-dose on Days 1,2,3 and 24 hours post last dose on Day 3 (Day 4)
Population: as for outcome 35
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanograms/milliliter
Arm/Group | Part B (10% BSA) GSK2646264 1% | Part B (3.5% BSA) GSK2646264 1%
Number analyzed (Participants) | 3 | 6
Hours*nanograms/milliliter
  Day 1, n=0, 0: number analyzed (Participants) | 0 | 0
  Day 2, n=0, 1: number analyzed (Participants) | 0 | 1
  Day 2, n=0, 1 |  | 34.4377 (NA) — NA indicates that geometric coefficient of variation could not be computed for Part B (3.5% BSA) GSK2646264 1% as a single participant was analyzed on Day 2.
  Day 3, n=3, 6 | 166.6914 (14) | 68.2224 (120)

49. Secondary Outcome: Area Under the Concentration-time Curve From Time 0 to Infinity (AUC [0-inf]) of GSK2646264 for Part B
Description: Blood samples were collected at the indicated time point to investigate the PK profile of GSK264624. From the GSK2646264 concentration-time data, the AUC (0-infinity) was determined using the currently approved and validated software.
Time Frame: Pre dose, 1 ,2, 4, 8, 12 hours post-dose on Days 1,2,3 and 24 hours post last dose on Day 3
Population: PK Population. Only those participants available at the indicated time points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*nanograms/milliliter
Arm/Group | Part B (10% BSA) GSK2646264 1% | Part B (3.5% BSA) GSK2646264 1%
Number analyzed (Participants) | 3 | 6
Hours*nanograms/milliliter
  Day 1: number analyzed (Participants) | 0 | 0
  Day 2: number analyzed (Participants) | 0 | 0
  Day 3 | 844.3091 (22) | 390.7973 (109)

50. Secondary Outcome: Terminal Half-life (t1/2) of GSK2646264 for Part B
Description: Blood samples were collected at the indicated time point to investigate the PK profile of GSK264624. From the GSK2646264 concentration-time data, the t1/2 was determined using the currently approved and validated software.
Time Frame: Pre dose, 1 ,2, 4, 8, 12 hours post-dose on Days 1,2,3 and 24 hours post last dose on Day 3
Population: PK Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Part B (10% BSA) GSK2646264 1% | Part B (3.5% BSA) GSK2646264 1%
Number analyzed (Participants) | 3 | 6
hours
  Day 1: number analyzed (Participants) | 0 | 0
  Day 2: number analyzed (Participants) | 0 | 0
  Day 3 | 59.69 (4.433) | 64.01 (11.220)

51. Secondary Outcome: Tmax of GSK2646264 for Part B
Description: as for outcome 43
Time Frame: Pre dose, 1 ,2, 4, 8, 12 hours post-dose on Days 1,2,3 and 24 hours post last dose on Day 3
Population: PK Population
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Part B (10% BSA) GSK2646264 1% | Part B (3.5% BSA) GSK2646264 1%
Number analyzed (Participants) | 3 | 6
hours
  Day 1 | 19.67 (23.6) | 17.85 (6.373)
  Day 2 | 16.93 (23.5) | 21.13 (6.436)
  Day 3 | 13.33 (24.0) | 12.62 (6.378)

52. Secondary Outcome: Cmax of GSK2646264 for Part C
Description: as for outcome 38
Time Frame: Pre dose and 4 hours post-dose on Days 1, 4 and 7
Population: PK Population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms/milliliter
Arm/Group | Part C GSK2646264 1%
Number analyzed (Participants) | 4
Nanograms/milliliter | 1.85336 (185)

53. Secondary Outcome: Tmax of GSK2646264 for Part C
Description: as for outcome 43
Time Frame: Pre dose and 4 hours post-dose on Days 1, 4 and 7
Population: PK Population
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Part C GSK2646264 1%
Number analyzed (Participants) | 4
hours | 4.10 (0.082)

54. Secondary Outcome: t1/2 of GSK2646264 for Part C
Description: Blood samples were collected at the indicated time point to investigate the PK profile of GSK264624. From the GSK2646264 concentration-time data, the t1/2 was determined using the currently approved and validated software. NA indicated data was not collected due to insufficient number of participants with data to calculate half life.
Time Frame: Pre dose and 4 hours post-dose on Days 1, 4 and 7
Population: PK Population
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Part C GSK2646264 1%
Number analyzed (Participants) | 4
hours | NA (NA) — NA indicated data was not collected due to insufficient number of participants with data to calculate half life.

ADVERSE EVENTS:
Time Frame: Non-serious AE and SAE were collected from Day 1 until follow-up (up to 11 days in Part A, 19 days in Part B and 23 days in Part C).
Description: Safety Population was used to collect AE and SAE.
Arm/Group | Part A-GSK2646264 0.5% | Part A-GSK2646264 1% | Part B (10% BSA)-Placebo | Part B (10% BSA) GSK2646264 1% | Part B (3.5% BSA)-Placebo | Part B (3.5% BSA) GSK2646264 1% | Part C-Placebo | Part C GSK2646264 1%
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/8 | 0/1 | 0/3 | 0/2 | 0/6 | 0/1 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/8 | 0/1 | 0/3 | 0/2 | 0/6 | 0/1 | 0/4
Other Adverse Events (participants affected / at risk) | 4/9 | 4/8 | 1/1 | 3/3 | 0/2 | 3/6 | 1/1 | 1/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A-GSK2646264 0.5% (N=9) | Part A-GSK2646264 1% (N=8) | Part B (10% BSA)-Placebo (N=1) | Part B (10% BSA) GSK2646264 1% (N=3) | Part B (3.5% BSA)-Placebo (N=2) | Part B (3.5% BSA) GSK2646264 1% (N=6) | Part C-Placebo (N=1) | Part C GSK2646264 1% (N=4)
Nasopharyngitis (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Application site erythema (General disorders) | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0
Application site pruritus (General disorders) | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1
Migraine (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pulpitis dental (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Skin test positive (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness postural (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2016-10-13): https://cdn.clinicaltrials.gov/large-docs/99/NCT02424799/Prot_000.pdf
  • Statistical Analysis Plan (2015-03-30): https://cdn.clinicaltrials.gov/large-docs/99/NCT02424799/SAP_001.pdf